CLINICAL TRIAL: NCT03903263
Title: Sleep Disturbances in Dermatology Patients- a Survey
Brief Title: Sleep Disturbances in Dermatology Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2018-00772; sp19Mueller
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorder
Keywords: dermatologic disease
MeSH Terms: conditions — Sleep Wake Disorders; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: survey on sleep disorders — self-administered patient questionnaire regarding the different aspects of sleep disorders in patients with dermatologic diseases

SUMMARY:
This study is to investigate sleep disorders in patients with dermatologic diseases by taking into consideration dermatologic (itch, pain) and non- dermatologic (medication, depression) factors.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of the dermatologic university clinic

Exclusion Criteria:

* Insufficient knowledge of German language
* Illiteracy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: outpatients of the dermatologic university clinic Basel
Sampling Method: Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Regensburg Insomnia Scale (RIS) | single time point assessment at baseline
  Self-rating scale: Five items cover quantitative and qualitative sleep parameters: Sleep latency (1), sleep duration (2), sleep continuity (3), early awakening (4) and sleep depth (5). Four items cover the psychological aspects of psychophysiological insomnia (PI), such as the experience of sleepless nights (6), focussing on sleep (7), fear of insomnia (8), and daytime fitness (9), one item covers sleep medication (10). A 5-step Likert scale was provided for response.The total score ranges from 0 to 40 points (score from 0-12 points considered as normal and a higher score as indicative of PI symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Müller, Dr. med, Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland